CLINICAL TRIAL: NCT07060443
Title: Clinico-oncological Safety and Efficacy of Real-time Fluorescence Lymph Node Mapping (FLNM) in Laparoscopic and Robotic Right Hemicolectomy for Patients With Locally Advanced Right-sided Colon Cancer; Multicenter Phase II Open Labelled Randomized Controlled Trial
Brief Title: Fluorescence Lymph Node Mapping for Colon Cancer Surgery
Acronym: CONSTELLARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Gyung Mo Son, Professor of Surgery, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-2024-001
Record Dates: First submitted 2025-05-22; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Right Hemicolectomy
MeSH Terms: interventions — Indocyanine Green; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLNM-guided Right Hemicolectomy (Experimental): FLNM-guided Right Hemicolectomy
  Interventions: Drug: Indocyanine green (ICG) injection for intraoperative lymph node imaging
- Right Hemicolectomy (Active Comparator): Standard Right Hemicolectomy without FLNM
  Interventions: Other: Standard Right Hemicolectomy (Non-ICG)

INTERVENTIONS:
Drug: Indocyanine green (ICG) injection for intraoperative lymph node imaging — Indocyanine Green (ICG) is used to guide the extent of D3 lymph node dissection during right hemicolectomy. After informed consent, participants randomized to the experimental group undergo bowel preparation and receive an endoscopic submucosal injection of ICG (0.25 mg/ml in saline) at two sites adjacent to the tumor one day prior to surgery. During surgery, near-infrared laparoscopic or robotic imaging systems detect the fluorescence emitted by ICG, guiding targeted D3 lymph node dissection at the origins of the ileocolic artery (ICA) and middle colic artery (MCA).
  Other Names: Fluorescence-guided Lymph Node Mapping
  Arms: FLNM-guided Right Hemicolectomy
Other: Standard Right Hemicolectomy (Non-ICG) — Participants in the control group undergo standard right hemicolectomy with D3 lymph node dissection without the use of Indocyanine Green (ICG) or fluorescence imaging. The extent of dissection is determined by conventional anatomical landmarks and the surgeon's clinical judgment.
  Other Names: Conventional Right Hemicolectomy
  Arms: Right Hemicolectomy

SUMMARY:
Fluorescence-guided surgery using indocyanine green can visualize the complex and diverse lymph node drainage structures for each patient and help determine the extent of dissection of the D3 lymph node tailored to the patient. However, since fluorescence lymph node mapping (FLNM) is still being conducted only at some institutions for research purposes and is limited to reporting the results of small-scale studies of patients, a large-scale multi-center study was conducted to verify the clinical-oncological effects of FLNM. Research is needed.

Therefore, this study used real-time fluorescence lymph node mapping (FLNM) to determine the extent of D3 lymph node dissection when performing right hemicolectomy and D3 lymph node dissection in patients with locally advanced right-sided colon cancer and to safely remove extensive lymph nodes. We aim to evaluate whether the dissection procedure is safe and beneficial in terms of clinical oncology.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who over 19 years old, Under 85 years old
2. Patient with locally advanced right colon cancer requiring D3 lymphadenectomy
3. Colon cancer patients diagnosed with clinical stage cT3-4 N0 or cTany N1-2 before surgery
4. Patient with right-sided colon cancer located in the cecum, ascending colon, flexure colon, and proximal transverse colon.
5. Patients with American Society of Anesthesiology (ASA) I-III
6. Patients who agreed to the research purpose and voluntarily gave informed consent

Exclusion Criteria:

1. Patients with a history of allergy or side effects to sodium iodine
2. Patients with colon cancer who have distant or peritoneal metastases
3. Patients requiring emergency surgery due to colon obstruction or colon perforation
4. Patients with inflammatory bowel disease not controlled by drug treatment
5. Patients with concurrent cancer in other areas other than colon cancer
6. Patients with a history of hereditary disease or coagulopathy at risk of bleeding
7. Women who are pregnant or may be pregnant and lactating women
8. Patients with chronic renal failure (e-GFR < 15) or patients receiving dialysis at the time of screening
9. Patients diagnosed with liver failure or with decreased consciousness due to hepatic encephalopathy
10. Patients judged to have difficulty in smooth lymph perfusion due to heart disease (acute myocardial infarction, acute and chronic heart failure) within the past 6 months
11. Patients unable to undergo general anesthesia
12. Patients with American Society of Anesthesiology (ASA) IV or V
13. Patients who do not wish to participate in this study
14. Patients who are judged by the researcher to be unsuitable for participation in this clinical trial (Example: People with a life expectancy of less than 6 months, people expected to have low compliance with clinical trials, etc.)

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-07-23 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological D3 lymph node metastasis detection rate | From enrollment to within 4 weeks after surgery

SECONDARY OUTCOMES:
Number of Harvest lymph nodes | From enrollment to within 4 weeks after surgery.
  Total lymph nodes, lymph nodes near tumor, D3 lymph nodes, ICA/RCA/MCA lymph nodes
Lymph Node Ratio (LNR) | From enrollment to within 4 weeks after surgery.
  LNR (lymph node ratio) = number of metastatic lymph nodes / total number of lymph nodes
Clinicopathological factors associated with FLNM success rate | From enrollment to within 8 weeks after surgery.
  Gender, age, BMI, pathological stage, tumor size, colon obstruction, etc
The bleeding rate due to damage to major blood vessels(SMA, SMV) during surgery | From enrollment to within 1 week after surgery.
Assessment of mesenteric dissection surface quality (3-point scale) | From enrollment to within 1 week after surgery
  A 3-point scoring system will be used to evaluate the quality of the mesenteric dissection surface following surgery. A higher score reflects a well-preserved mesenteric dissection surface with minimal or no damage.
  * 3 points: Complete mesenteric dissection (the dissection surface is intact, with no visible damage, and the peritoneal surface is well preserved)
  * 2 points: Nearly complete mesenteric dissection (the dissection surface shows some damage, but there is no exposure of tumor tissue)
  * 1 point: Incomplete mesenteric dissection (the dissection surface is damaged, with exposure of tumor tissue within the colonic wall.)
Proximal and distal lengths(cm) | From enrollment to within 1 week after surgery
  Proximal and distal resection lengths
Estimated Blood loss(ml) | On the day of surgery
Operation time(min) | On the day of surgery
Complications | Within 30 days after surgery
  This outcome measure assesses postoperative complications occurring within 30 days after surgery. Complications are classified according to the Clavien-Dindo classification system, which grades adverse events based on their severity and the type of intervention required. Trained clinical staff will record and categorize complications during the postoperative follow-up period.
Readmission | Within 30 Days After Surgery
  This outcome measure records whether patients are readmitted to the hospital within 30 days after surgery. In cases of readmission, the reason for readmission will be documented, including complications, treatment-related issues, or other causes as determined by clinical evaluation.
Reoperation | Within 30 Days After Surgery
  This outcome measure records whether patients undergo reoperation within 30 days after the initial surgery. The reasons for reoperation, such as complications or surgical site issues, will be documented based on clinical evaluation.
Completeness score of D3 lymph node dissection (3-point scale) | Assessed on the day of surgery
  A 3-point scoring system will be used intraoperatively to assess the completeness of D3 lymph node dissection using real-time fluorescence imaging.
  Higher scores indicate a more complete lymph node dissection.
  * 1 point: Residual fluorescent lymph nodes are present in the D3 area (justification required).
  * 2 points: Residual fluorescent lymph nodes are present but resection is deemed unnecessary by the surgeon (e.g., outside D3 area; justification required).
  * 3 points: No residual fluorescent lymph nodes remain in the D3 area.
3year disease-free survival rate | From enrollment to 3 years after surgery
overall survival rate | From enrollment to 5 years after surgery
local and systemic recurrence rate | From enrollment to 3 years after surgery
Surgeon perceptions of FLNM-guided D3 lymphadenectomy | - Before enrollment of the first subject (after IRB approval) - At the end of enrollment of all subjects
  * A custom survey developed by the research team will assess surgeons' perceptions of the usefulness, safety, and potential future application of Fluorescence lymph node mapping (FLNM) guided D3 lymphadenectomy in colorectal cancer surgery. The survey includes Likert-type questions (e.g., "Strongly agree" to "Strongly disagree") and multiple-choice items (e.g., "For which patients is FLNM used?").
  * Responses will be reported as the proportion of participants selecting each option for key questions, such as:
    * Is FLNM helpful for determining the lymph node dissection range?
    * Do you plan to use FLNM in future surgeries?
    * Do you believe FLNM helps reduce complications?
    * For which patient groups is FLNM currently used?
  * The survey will be conducted at two time points: (1) before enrollment of the first subject (after IRB approval), and (2) after enrollment of all subjects has been completed.

CONTACTS AND LOCATIONS:
Locations (13):
- South Korea (13):
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center Korea, Goyang
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil Medical Center, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No